CLINICAL TRIAL: NCT00976196
Title: Platelet Hyperreactivity Project: A System Biology Approach of High On-treatment Platelet Reactivity in Aspirin-treated Cardiovascular Patients
Brief Title: Platelet Hyperreactivity Project
Acronym: PHP
Status: Completed | Type: Observational
Sponsor: Pierre Fontana (Other)
Responsible Party: Sponsor-Investigator, Pierre Fontana, PI, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 08-104
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Platelet Reactivity
Keywords: Aspirin; Blood platelets; proteomics; Platelet reactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Serum Platelets
Oversight: Data Monitoring Committee: No

SUMMARY:
The PHP study aims to delineate gene products involved in high on-treatment platelet reactivity in aspirin-treated cardiovascular patients.

DETAILED DESCRIPTION:
The PHP study aims to delineate gene products involved in high on-treatment platelet reactivity in aspirin-treated cardiovascular patients using a system biology approach that include proteomics analysis of selected platelet sub-fractions in patients displaying extreme phenotype.

Main objective:

* to characterize the proteome profile of platelet hyperreactivity in aspirin-treated cardiovascular patients

Secondary objectives:

* to characterize the platelet hyperreactivity phenotype in cardiovascular patients treated with aspirin
* to determine genetic polymorphisms associated with platelet hyperreactivity

ELIGIBILITY:
Inclusion Criteria:

* Documented symptomatic ischemic atherothrombotic disease treated by aspirin.

Exclusion Criteria:

* Known platelet disorder
* Chronic treatment by antiplatelet drugs other than aspirin
* Chronic anticoagulant treatment
* Chronic non steroidal anti-inflammatory drug treatment
* Active cancer
* Treatment with serotonin reuptake inhibitors

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic atherothrombotic patients treated with aspirin.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
proteome profile of platelet hyperreactivity | cross sectional
  to characterize the proteome profile of platelet hyperreactivity in aspirin-treated cardiovascular patients

SECONDARY OUTCOMES:
platelet hyperreactivity phenotype in cardiovascular patients treated with aspirin | cross sectional

OTHER OUTCOMES:
genetic polymorphisms associated with platelet hyperreactivity | cross sectional

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fontana, MD, PhD, Principal Investigator — University of Geneva
Locations (1):
- University Hospital Geneva, Geneva, Switzerland